CLINICAL TRIAL: NCT02417506
Title: A Double Blind Randomized Comparator Controlled Study to Assess the Effect of E-OA-07 (Lanconone) on Acute Pain Response in Subjects Suffering From Osteoarthritis of the Knee
Brief Title: Study to Assess the Effect of E-OA-07 on Acute Pain Response in Subjects Suffering From Knee OA
Acronym: Osteolanc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Enovate Biolife Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EB/ 140501 /LC/ OA
Record Dates: First submitted 2015-01-21; First posted 2015-04-15 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis of Knee
Keywords: Acute pain; Herbal; VAS; Stop watch
MeSH Terms: conditions — Osteoarthritis, Knee; Acute Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-OA-07 (Lanconone) (Experimental): 500 mg two capsules to be taken stat at the site
  Interventions: Other: E-OA-07 (Lanconone)
- Ibuprofen (Active Comparator): 200 mg two capsule to be taken stat at the site
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Other: E-OA-07 (Lanconone)
  Other Names: Investigational Product
  Arms: E-OA-07 (Lanconone)
Drug: Ibuprofen
  Other Names: Comparator
  Arms: Ibuprofen

SUMMARY:
The repetitive motions associated with active life and many sports can increase the wear and tear to the joints that leads to decrease in flexibility and joint pain finally heading its way to osteoarthritis. Activities such as jumping, running can wear away the cartilage that supports and cushions the joints of hands and knees, causing bones to rub against each other. Injuries stemming from repetitive motions can also cause and worsen the joint pain.

Joint pain is discomfort that arises from any joint . Irrespective of the underlying mechanisms, joint pain usually originates in activation of nociceptors, or free nerve endings. Complex neuronal activation occurs, which involves not only local sensitization of joint nociceptors but also modifications in central pain pathways.

Even though, the numerous pharmacological interventions are available for joint pain, there is much debate amongst clinicians about the best approach to the treatment of joint pain. NSAIDs which is frequently used for treatment in such cases, carries concerns related to gastro-intestinal system, cardiovascular system as well as central nervous system .

Hence there is a need of a safer alternative treatment option for relieving acute joint pain which is comparable to the modern medicines, without posing concerns to the subject's general well being.

Herbs are known to be used since ages in traditional literature and do not pose any potential health concern. Inspite of such positive attributes herbs are not employed in treatment of acute pains as there is lack of evidence proving the same.

In order to address the need of the hour Enovate Biolife has invented a novel poly herbal formulation E-OA-07 (Lanconone). Lanconone has been studied previously in patients with osteoarthritis has been proven efficacious . It has a good history of marketing and is sold in the United States, with no reported adverse event related to the product. However there is no concrete evidence proving the product's acute pain relieving dynamics, hence the current study has been employed to comprehend the effect of lanconone in joint acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adults of either sex aged 40 to 60 years.
* Subjects with moderate OA of the knee, which can be clinically, categorized as ARA functional Class II and III with radiological confirmation of Kellgren Lawrence Grade II and III. (incase of bilateral OA, the knee with the more severe symptoms will be defined as index joint)
* Subjects with OA in a flare state at the baseline defined by one of following category of flare:

In subjects who have been receiving non steroidal anti-inflammatory drugs (NSAIDs) or analgesic therapy for their OA, flare will be defined as having at least two of the following three criteria while comparing screening to baseline:

1. Subject's assessment of arthritis pain VAS walking on a flat surface at baseline of ≥ 40 mm;
2. Increase of ≥ 1 grade in the patients global assessment of arthritis;
3. Increase of ≥ 1 grade in the physician's global assessment of arthritis;

In subjects who are not receiving NSAID or analgesic therapy , an OA flare state will be defined as having at least two of the following three criteria

1. Subject's assessment of arthritis pain VAS walking on a flat surface at baseline of ≥ 40 mm
2. Patient's global assessment of arthritis of ''poor''; very poor
3. Physician's global assessment of arthritis of ''poor''; very poor

Exclusion Criteria:

* Subjects with any form of arthritis other than osteoarthritis.
* Administration of intra-articular or oral steroids in the past 3 month or intra articular hyaluronic acid in the last 9 months or parenteral use of NSAIDs
* History of major chronic hepatic, cardiovascular, neurological or immunosuppressive conditions or the presence of any infections
* Subjects with localized trauma to the lower limb
* Had received oral, intramuscular, or intra-articular corticosteroids within 8 weeks, or intra-articular hyaluronic acid in the index joint within 6 months of study drug administration;
* Subjects on nutritional supplement or herbal product since last one month
* Subjects otherwise judged by the investigator to be inappropriate for inclusion in the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pain score as measured by Visual Analogue Scale | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Srivastava, M.D., Study Chair
Locations (1):
- Mukund Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Girandola RN, Srivastava S, Loullis CC. A clinical trial comparing Lanconone(R) with ibuprofen for rapid relief in acute joint pain. Trials. 2016 Apr 6;17:189. doi: 10.1186/s13063-016-1268-6. PMID 27052991